CLINICAL TRIAL: NCT04380883
Title: Combination of InnoSEAL Plus TR Band Compared to TR Band Alone for Radial Artery Outcomes in Patients Undergoing Transradial Coronary Intervention (InnoSEAL II)
Brief Title: Combination of InnoSEAL Plus TR Band Compared to TR Band Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tabba Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InnoSEAL II
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Radial Artery Occlusion; Hematoma
Keywords: radial artery occlusion; access site outcomes; hemostatic patch
MeSH Terms: conditions — Arterial Occlusive Diseases; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- InnoSEAL+TRB (Experimental): InnoSEAL is a hemostatic patch which will be applied along with TRB to control bleeding from access site
  Interventions: Device: InnoSEAL+TRB
- TRB alone (Active Comparator)
  Interventions: Device: TRB alone

INTERVENTIONS:
Device: InnoSEAL+TRB — InnoSEAL is a catecholamine chitosan-based pad (InnoSEAL hemostatic pad, InnoTherapy, Inc.). Chitosan-Catechol in InnoSEAL instantly forms an adhesive barrier upon blood contact. It is intended for use under the care of a healthcare professional. The dressing is indicated for the skin surface puncture sites for vascular procedures, percutaneous catheters/tubes. TRB is a pneumatic device which is applied routinely at the puncture site and inflated with air to stop bleeding from the access site. We will apply InnoSEAL and TRB together.
  Arms: InnoSEAL+TRB
Device: TRB alone — TRB is a pneumatic device which is applied routinely at the puncture site and inflated with air to stop bleeding from the access site. It will be the comparing arm.
  Arms: TRB alone

SUMMARY:
Angiography or angioplasty are commonly now done through inserting the device through radial artery in hand i.e. trans-radial procedures. It is reported that between 2-30% of these procedures get complicated by radial artery occlusion (RAO) which limit future use of this site for similar procedures if needed. It is important to control the arterial bleeding after the procedure completion while maintaining radial arterial flow appears to be an important factor in reducing RAO (patent hemostasis). Currently the most frequently employed method for hemostasis following trans-radial procedures is a compression device (RCD) such as TransRadial Bands (TRB). But TRB takes hours to achieve hemostasis and causes discomfort to the patients and longer time to discharge. Hemostatic pads offer an alternative to RCD where overall compression time is inherently low and patent hemostasis can possibly be achieved. The combined use of TR band with a hemostatic device may allow ease of use with reduced hemostasis time.

The trial aims to test the hypothesis that compared to TR band (TRB) alone, catecholamine chitosan-based pad (InnoSEAL hemostatic pad, InnoTherapy, Inc.) used in conjunction with TRB (InnoSEAL+TRB)is nearly as good as TRB alone in terms of the outcomes like RAO and hematoma.

DETAILED DESCRIPTION:
It is a prospective, randomized, open label trial with the following study hypotheses (Ha):

1. InnoSEAL+TRB is non-inferior to TRB alone in terms of the composite adverse access site outcomes including RAO and hematoma.
2. InnoSEAL+TRBis non-inferior to TRB alone when comparing ease of use scores rated by the cath lab technicians.
3. InnoSEAL+TRB is superior to TRB alone for outcomes of reduction in total hemostasis time, total observation time for the radial site and time to hospital discharge for daycare patients sub group.
4. InnoSEAL+TRBis superior to TRB alone in terms of minimized patient discomfort.

Sample size:

Keeping a combined complication rate of 17.7% (RAO:7.7%, Hematoma: 10%), difference in favor of the experimental treatment of 4.89%, power of 80%, one sided alpha of 2.5%, 10% attrition rate, a sample of at least 357 patients in each group and a total of 714 patients will be required.

Randomization:

Randomization will be performed using variable sized blocks through computer software by an unrelated staff from the research department who is not a part of this study and will be kept in safe in the research department. Allocation of intervention will be informed to the research staff for each individual patient through telephone call, only after the informed consent has been taken by the data collector.

Intervention arm:

In InnoSEAL+TRB arm, InnoSEAL patch will be applied at the puncture site and will be covered by a transparent dressing. TRB will be applied over the patch and 12 cc air will be injected to inflate the band. Air is removed from TRB during 60 minutes, removing 2cc air at 20 minutes, 4cc at 40 minutes and 6cc at 60 minutes from the time of sheath removal.

Control arm:

TR band is applied centered over the puncture site and the bladder is inflated with 15cc air. Air is removed gradually leaving at least 10 cc air provided there is no oozing. Start removing air at 90 min (from the time of hemostasis protocol):

4cc-at 20 min, 6cc-at 40 min. 6cc-at each 20 min till reach 0cc. If re-bleeding at any time, reintroduce 2cc air.

In both the arms TRB will be left with 0cc air for 30 min. Reverse Barbeau's test will be applied in both the arms to determine RAO. If occlusion was found, radial artery ultrasound will be conducted. Both TRB and InnoSEAL patch will be removed before discharge of the patient.

Data quality measures:

Data will be collected by the trained nursing staff hired specifically for the study and who will receive one day training on study protocols. Study coordinator will daily check all the forms for completeness and accuracy and 10% of the completed forms will be randomly checked by one of the study investigators. Institutional IRB will also do an audit of the study procedures.

Data entry and analysis:

Data will be entered in Access data base and will be analyzed through SPSS v.25. Means and standard deviation will be reported for continuous data based on normality assumption along with histograms and compared using Student t-test. And frequencies with percentages will be reported for the categorical variables. The differences between categorical variables were examined by the Chi square test considering p-value< .05 statistically significant. Chi square test will be utilized to assess primary composite outcome and its components. Independent sample t-test will be used for comparison of time intervals. Kruskall Wallis test will be utilized for significance testing between ordinal secondary outcomes of ease of use and patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both gender undergoing coronary procedure using trans radial approach (diagnostic or PCI) will be included
* Both elective and hemodynamically stable, acute coronary syndrome (ACS) patients will be included.

Exclusion Criteria:

* Sheath larger than 6F
* IV Heparin or GP 2b/3a inhibitors continued after the procedure
* Ongoing anticoagulation with Warfarin or Rivaroxaban or INR > 3
* Ipsilateral AV fistula
* Barbeau's Class D
* History of RAO at baseline
* Patients unable to give consent due to clinical instability or sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Access site combined outcomes | within 24 hours
  Proportion of patients with RAO and/or hematoma of any grade.
  1. Radial artery occlusion: Radial artery will be defined as occluded if reverse Barbeau's test shows absence of flow on pulse oximetry just after the removal of the TR band in both groups.In patients identified to have RAO, findings will be confirmed using UltraSound (US) Duplex using color flow with pulse wave imaging within 24 hours of the radial procedure.US Duplex will be performed during the index hospital stay.
  2. Radial Hematoma: Radial artery site will be assessed for presence of hematoma at the end of hemostasis protocol. Hematoma will be marked if present, and graded according to categories of I-IV. Hematomas grade II-IV will be considered significant.

SECONDARY OUTCOMES:
Ease of use | Upto 30 weeks
  Ease of use of InnoSEAL will be assessed by a system usability scale (SUS), 5 point Likert scale by the cath lab personnel who routinely perform post procedure hemostasis. Ease of use is reported as percentage acceptability where 100% means highly acceptable and vice versa. Ease of use proforma will be filled by the participating cath lab staffs at the end of the study.
Total compression time: | within 24 hours
  Time required from radial sheath removal to the removal of all the air from TR band.
Total observation time: | within 24 hours
  Time required from radial sheath removal to the removal of TR band (included time for observation at 0 cc for safety purpose).
Time to hospital discharge: (For daycare patients only) | within 24 hours
  Time from removal of radial sheath till patient discharge from hospital
Patient discomfort: | within 24 hours
  Standard visual pain scale of 1-10 will be utilized. Pain will be assessed after the hemostasis protocol is ended.

CONTACTS AND LOCATIONS:
Locations (1):
- Tabba Heart Institute, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Aijaz S, Sheikh S, Pathan A. Combination of InnoSEAL plus TR band compared with TR band alone for radial artery outcomes in patients undergoing transradial coronary intervention (InnoSEAL-II): an open-label randomised controlled trial (protocol). BMJ Open. 2020 Dec 23;10(12):e042101. doi: 10.1136/bmjopen-2020-042101. PMID 33361166